CLINICAL TRIAL: NCT04279054
Title: Decreased Neuraxial Morphine and Adjunctive Peripheral Nerve Blockade to Reduce Severity of Side Effects and Opioid Use After Cesarean Delivery
Brief Title: Decreased Neuraxial Morphine After Cesarean Delivery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ayodeji Sanusi, Principal Investigator/ Assistant Professor Maternal Fetal Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00000196; UL1TR003096 (NIH)
Record Dates: First submitted 2020-02-13; First posted 2020-02-20 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia
Keywords: cesarean delivery; epidural; Neuraxial block; anesthesia side effects
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A: 150 mcg morphine (Active Comparator): Patients in this group will receive 150mcg of morphine in their neuraxial block
  Interventions: Drug: Morphine Sulfate 150 mcg
- Group B: 50 mcg morphine (Experimental): Patients in this group will receive 50mcg of morphine in their neuraxial block
  Interventions: Drug: Morphine Sulfate 50mcg

INTERVENTIONS:
Drug: Morphine Sulfate 150 mcg — Use of 150mcg of morphine sulfate for neuraxial block (dosing difference)
  Arms: Group A: 150 mcg morphine
Drug: Morphine Sulfate 50mcg — Use of 50mcg of morphine sulfate for neuraxial block (dosing difference)
  Arms: Group B: 50 mcg morphine

SUMMARY:
The purpose of this study is to compare 50mcg to 150mcg morphine in epidural for the goal of decreasing side effects of medication with lower dose in patients who receive a QL block

DETAILED DESCRIPTION:
Regional anesthesia has been associated with reduced opioid consumption after surgery. Cesarean delivery is one of the most commonly performed surgeries worldwide and women undergoing cesarean delivery are often young, opioid-naïve, and motivated to recover quickly in an effort to better care for their newborn. However, approximately 1 in 300 opioid naïve women become persistent prescription opioid users following cesarean delivery . Hence, it is important to optimize post-cesarean pain control while limiting exposure to opioids. Currently, standard therapy includes the use of neuraxial morphine (NM) in combination with a multi-modal regime in an effort to limit excessive opioid use after cesarean delivery. The current typical dose of NM that is given prior to cesarean delivery at the investigator's center is 150 mcg. Importantly, NM doses as low as 100 mcg have been shown to provide comparable analgesia while reducing side effects such as itching. The side-effect profile associated with NM includes up to 87% of patients experiencing pruritus and up to 70% experiencing urinary retention. Nausea and vomiting also lead to significant discomfort for a new mother trying to provide acute infant care.

Adjunctive Peripheral Nerve Blockade has recently been introduced to reduce postoperative pain and opioid use. Studies have assessed the usefulness of the transversus abdmoninis plane (TAP) block after cesarean delivery. Another ultrasound-guided injection of local anesthetic in the fascial plane (truncal block) that is available at UAB and within the standard of care for patients undergoing abdominal surgery is the quadratus lumborum (QL) block. Because of its more posterior and caudal location, it is more likely to anesthetize the nerve fibers associated with pain from cesarean delivery.

This study will compare the use of 50mcg to 150mcg morphine for the goal of decreasing side effects of medication with lower dose in all patients who receive a QL block

ELIGIBILITY:
Inclusion Criteria:

* All women presenting for scheduled cesarean delivery who desire a QL block

Exclusion Criteria:

* Women with pregnancies complicated by preeclampsia
* Women with pregnancies complicated by insulin-treated diabetes
* Women with pregnancies complicated by placental abnormalities
* Women with pregnancies complicated by a history of opioid use disorder

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Outcome of side effects of intervention: pruritus | One assessment during hospital stay - up to postoperative day 2 (2 days following cesarean delivery)
  Incidence of primary outcome surrogate marker by need for medication for pruritus based on verbal complaints from patient (Medication given: Yes or No)
Outcome of side effects of intervention: nausea | One assessment during hospital stay - up to postoperative day 2
  Incidence of primary outcome surrogate marker by need for medication for nausea based on verbal complaints from patient (Medication given: Yes or No)
Outcome of side effects of intervention: urinary retention | One assessment during hospital stay - up to postoperative day 2 (2 days following cesarean delivery)
  Incidence of primary outcome surrogate marker by need for removal of foley catheter as measure for urinary retention

SECONDARY OUTCOMES:
Maternal secondary outcomes from intervention | One assessment during hospital stay - up to postoperative day 2 (2 days following cesarean delivery)
  Total amount of morphine use during hospital stay (cumulative morphine administered to control pain during hospital stay)
Maternal secondary outcomes from intervention | One measurement during entire hospital stay
  Incidence of daily pain scores (measured by pain score ratings: 1-10); 1: lowest pain score 10: maximum pain score
Neonatal secondary outcomes from intervention | Within first hour of birth
  Apgar scores
Neonatal secondary outcomes from intervention | Within first hour of birth
  Incidence of babies with signs of respiratory depression

CONTACTS AND LOCATIONS:
Overall Officials: Ayodeji Sanusi, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Women and Infants Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donauer K, Bomberg H, Wagenpfeil S, Volk T, Meissner W, Wolf A. Regional vs. General Anesthesia for Total Knee and Hip Replacement: An Analysis of Postoperative Pain Perception from the International PAIN OUT Registry. Pain Pract. 2018 Nov;18(8):1036-1047. doi: 10.1111/papr.12708. Epub 2018 Jun 25. PMID 29758587
- [Background] Bateman BT, Franklin JM, Bykov K, Avorn J, Shrank WH, Brennan TA, Landon JE, Rathmell JP, Huybrechts KF, Fischer MA, Choudhry NK. Persistent opioid use following cesarean delivery: patterns and predictors among opioid-naive women. Am J Obstet Gynecol. 2016 Sep;215(3):353.e1-353.e18. doi: 10.1016/j.ajog.2016.03.016. Epub 2016 Mar 17. PMID 26996986
- [Background] Girgin NK, Gurbet A, Turker G, Aksu H, Gulhan N. Intrathecal morphine in anesthesia for cesarean delivery: dose-response relationship for combinations of low-dose intrathecal morphine and spinal bupivacaine. J Clin Anesth. 2008 May;20(3):180-5. doi: 10.1016/j.jclinane.2007.07.010. PMID 18502360
- [Background] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500
- [Background] McDonnell JG, Curley G, Carney J, Benton A, Costello J, Maharaj CH, Laffey JG. The analgesic efficacy of transversus abdominis plane block after cesarean delivery: a randomized controlled trial. Anesth Analg. 2008 Jan;106(1):186-91, table of contents. doi: 10.1213/01.ane.0000290294.64090.f3. PMID 18165577
- [Background] McMorrow RC, Ni Mhuircheartaigh RJ, Ahmed KA, Aslani A, Ng SC, Conrick-Martin I, Dowling JJ, Gaffney A, Loughrey JP, McCaul CL. Comparison of transversus abdominis plane block vs spinal morphine for pain relief after Caesarean section. Br J Anaesth. 2011 May;106(5):706-12. doi: 10.1093/bja/aer061. PMID 21498494
- [Background] Faiz SHR, Alebouyeh MR, Derakhshan P, Imani F, Rahimzadeh P, Ghaderi Ashtiani M. Comparison of ultrasound-guided posterior transversus abdominis plane block and lateral transversus abdominis plane block for postoperative pain management in patients undergoing cesarean section: a randomized double-blind clinical trial study. J Pain Res. 2017 Dec 19;11:5-9. doi: 10.2147/JPR.S146970. eCollection 2018. PMID 29296094
- [Background] Champaneria R, Shah L, Wilson MJ, Daniels JP. Clinical effectiveness of transversus abdominis plane (TAP) blocks for pain relief after caesarean section: a meta-analysis. Int J Obstet Anesth. 2016 Dec;28:45-60. doi: 10.1016/j.ijoa.2016.07.009. Epub 2016 Aug 5. PMID 27717634
- [Background] Ng SC, Habib AS, Sodha S, Carvalho B, Sultan P. High-dose versus low-dose local anaesthetic for transversus abdominis plane block post-Caesarean delivery analgesia: a meta-analysis. Br J Anaesth. 2018 Feb;120(2):252-263. doi: 10.1016/j.bja.2017.11.084. Epub 2017 Dec 5. PMID 29406174
- [Background] Quinlan JD, Murphy NJ. Cesarean delivery: counseling issues and complication management. Am Fam Physician. 2015 Feb 1;91(3):178-84. PMID 25822271
- [Background] Lavand'homme P. Postcesarean analgesia: effective strategies and association with chronic pain. Curr Opin Anaesthesiol. 2006 Jun;19(3):244-8. doi: 10.1097/01.aco.0000192815.22989.61. PMID 16735805
- [Background] Committee Opinion No. 666: Optimizing Postpartum Care. Obstet Gynecol. 2016 Jun;127(6):e187-e192. doi: 10.1097/AOG.0000000000001487. PMID 27214194
- [Background] Abdallah FW, Laffey JG, Halpern SH, Brull R. Duration of analgesic effectiveness after the posterior and lateral transversus abdominis plane block techniques for transverse lower abdominal incisions: a meta-analysis. Br J Anaesth. 2013 Nov;111(5):721-35. doi: 10.1093/bja/aet214. Epub 2013 Jun 27. PMID 23811424
- [Background] Telnes A, Skogvoll E, Lonnee H. Transversus abdominis plane block vs. wound infiltration in Caesarean section: a randomised controlled trial. Acta Anaesthesiol Scand. 2015 Apr;59(4):496-504. doi: 10.1111/aas.12498. PMID 25786679
- [Background] Blanco R, Ansari T, Riad W, Shetty N. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Pain After Cesarean Delivery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):757-762. doi: 10.1097/AAP.0000000000000495. PMID 27755488
- [Background] Hirabayashi M, Doi K, Imamachi N, Kishimoto T, Saito Y. Prophylactic Pentazocine Reduces the Incidence of Pruritus After Cesarean Delivery Under Spinal Anesthesia With Opioids: A Prospective Randomized Clinical Trial. Anesth Analg. 2017 Jun;124(6):1930-1934. doi: 10.1213/ANE.0000000000002060. PMID 28448397
- [Background] Aly M, Ibrahim A, Farrag W, Abdelsalam K, Mohamed H, Tawfik A. Pruritus after intrathecal morphine for cesarean delivery: incidence, severity and its relation to serum serotonin level. Int J Obstet Anesth. 2018 Aug;35:52-56. doi: 10.1016/j.ijoa.2018.02.004. Epub 2018 Feb 16. PMID 29544720